CLINICAL TRIAL: NCT01231204
Title: Prevention of Post-Mastectomy Breast Pain Using Ambulatory Continuous Paravertebral Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVB Catheter Study
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Paravertebral Catheter Insertion; Mastectomy; Breast Cancer
Keywords: Breast Cancer; Mastectomy; UCSD; Surgery; PVB Catheter; Paravertebral Catheter; Breast Pain; Mastectomy Pain; Postoperative Pain
MeSH Terms: conditions — Breast Neoplasms; Mastodynia; Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Infusion (Placebo Comparator): Patients will be randomized to receive a continuous infusion of Normal Saline via a Paravertebral Nerve Block.
  Interventions: Procedure: Placebo (normal saline) Continuous Infusion
- Ropivicaine 0.4% Infusion (Active Comparator): Patients will be randomized to receive a continuous infusion of 0.4% Ropivicaine via a Paravertebral Nerve Block.
  Interventions: Procedure: Ropivicaine 0.4% Continuous Infusion

INTERVENTIONS:
Procedure: Placebo (normal saline) Continuous Infusion — Patients randomized to this group will receive an initial catheter placement using the standard Ultrasound-guided Technique. For the surgical procedure they will receive 15cc of 0.5%Ropivicaine. Following the surgical procedure they will receive a pain pump filled with normal saline. The normal saline infusion will continue for the 3 days following surgery. All patients will have access to other pain relievers for break-through pain. All patients will have the outcome measures assessed.
  Arms: Placebo Infusion
Procedure: Ropivicaine 0.4% Continuous Infusion — Patients randomized to this group will receive an initial catheter placement using the standard Ultrasound-guided Technique. For the surgical procedure they will receive 15cc of 0.5%Ropivicaine. Following the surgical procedure they will receive a pain pump filled with 0.4%Ropivicaine. The 0.4%Ropivicaine infusion will continue for the 3 days following surgery. All patients will have access to other pain relievers for break-through pain. All patients will have the outcome measures assessed.
  Arms: Ropivicaine 0.4% Infusion

SUMMARY:
Research study to determine if putting local anesthetic-or numbing medication-through a tiny tube placed next to the nerves that go to a breast prior to and following a mastectomy will decrease subsequent pain.

DETAILED DESCRIPTION:
Specific Aim 1: To determine if, compared with current and customary analgesia, the addition of a multiple-day ambulatory continuous paravertebral block decreases the incidence and severity of post-mastectomy pain.

Hypothesis 1: Following mastectomy, the incidence and severity of breast pain will be significantly decreased in the week following surgery with a multiple-day ambulatory continuous paravertebral block as compared with patients receiving standard-of-care treatment (as measured on the 11-point numeric rating scale).

Hypothesis 2: Following mastectomy, the incidence and severity of chronic pain will be significantly decreased three months following multiple-day ambulatory continuous paravertebral blocks as compared with patients receiving standard-of-care treatment (as measured on the 11-point numeric rating scale).

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral or bilateral mastectomy
* desiring analgesia with a paravertebral nerve block(s)
* age 18 years or older
* female

Exclusion Criteria:

* morbid obesity as defined by a body mass index > 40
* renal insufficiency
* chronic opioid use
* history of opioid abuse
* any comorbidity which results in moderate or severe functional limitation
* inability to communicate with the investigators or hospital staff
* pregnancy
* incarceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pain Scores (NRS) | Day following Surgery
  Pain score on the 0-10 Numeric Rating Scale given as part of the Brief Pain Inventory

SECONDARY OUTCOMES:
Pain scores | First 4 postoperative days
  Measured on the NRS (defined above) during the first 4 postoperative days
Opioid Requirements | First 4 postoperative days
  Both in and out of the hospital during the first 3 postoperative days
Opioid-related side effects | First 4 postoperative days
  Both in and out of the hospital during the first 4 postoperative days
Sleep Disturbances | First 4 postoperative days
  Due to breast pain during the first 4 postoperative days
Cancer Recurrence | One Year following Surgery
  Patients' records will be investigated for indications of cancer recurrence up to 3 years following catheter placement (including estrogen receptor status as + or -). Patients may be contacted by phone if records suggest that the patient has not returned to the original surgeon within the previous 12 months
Pain and Physical Functioning | Within first year of surgery
  Brief Pain Inventory given by phone on postop day 1, 4, 8; and weeks 4, 12; and months 3 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego, Department of Anesthesia
Locations (1):
- UCSD Thornton Hospital, La Jolla, California, United States